CLINICAL TRIAL: NCT02957773
Title: Integration of Social Art Activities and Qigong Exercises to Increase the Well-Being of Older People in Nursing Homes in Indonesia
Brief Title: Integration of Social Art Activities and Qigong for Older People in Nursing Home in Indonesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Universitas Tarumanagara (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SAAQE-R053
Record Dates: First submitted 2016-09-28; First posted 2016-11-08 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2016-09

CONDITIONS: Well-being; Depressive Symptoms
MeSH Terms: conditions — Depression | interventions — Qigong; Activities of Daily Living

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Qigong and art activities (Experimental): An integrated group of Qigong and art activities for 90 minutes.
  Interventions: Behavioral: Qigong and art activities
- Art activities (Experimental): Art activities and daily activities group for 90 minutes.
  Interventions: Behavioral: Art activities
- Qigong (Experimental): A Qigong and daily activities group for 90 minutes
  Interventions: Behavioral: Qigong
- Daily activities (Other): A daily activities group for 90-minutes.
  Interventions: Behavioral: Daily activities

INTERVENTIONS:
Behavioral: Qigong and art activities — Participants join a 90-minute session of integrated Qigong and art activity consisting of 30 minutes Qigong followed by 60 minutes art activity.
  Arms: Qigong and art activities
Behavioral: Art activities — Participants join a 90-minute session that consists of 60-minute art activities followed by 30 minutes daily activities.
  Arms: Art activities
Behavioral: Qigong — Participants join a 90-minute session that consists of 30-minutes Qigong exercise followed by 60 minutes daily activities (watching television, reading or sitting together).
  Arms: Qigong
Behavioral: Daily activities — Participants do their daily activities routine for 90-minutes, such as watching television, reading and sitting together or participants can do free individual activities on their own.
  Arms: Daily activities

SUMMARY:
This project will be a randomised controlled trial to investigate the effectiveness of an integrated programme by using social art activity (SA) and exercise, for instance, Qigong (QG, a traditional Chinese exercise) as a therapeutic medium.

This integrated programme aims to increase the well-being and reduce the depressive symptoms that are frequently ascertained in older people who live in nursing homes. The combination of SA and QG might be more beneficial to older people than either individual activity on its own, given that they are addressing different areas of functioning. The art activity focuses on self-expression in non-verbal activity using fine motor movement, whereas physical exercise like Qigong focuses on awareness of breathing and a calm state of mind. This is to help the older person achieve mental and physical relaxation by using gross motor movement. When the interventions are combined by utilising Qigong ahead of the art activities (thus, including both fine and gross motor movements) older people will reach a state of mental and physical relaxation, and moreover, will be able to express their feelings more simply in the social art activities.

DETAILED DESCRIPTION:
Depression is one of the most common mental disorders with regards to older people. It is a serious disease affecting an individual's entire life-situation, which can lead to suffering and a reduced level of activity in everyday life. Depression inhibits thinking capacity in self-expression and reduces the ability to communicate. Furthermore, older people with depression often use a considerable amount of energy attempting to avoid distressing emotions and negative thinking, which is one of the principal symptoms of depression.

Research findings describing the use of relaxation or meditation to prepare clients prior to the art activities are effective treatment methods in the reduction of depression and anxiety. However, adding Qigong as an initial therapy prior to the art activities enhances the effectiveness of art therapy. When older people achieve deep states of mental and physical relaxation, they will be able to activate their thinking capacity regarding self-expression by means of the use of art media. Thus, their negative feelings will be directed toward art activities, which in turn will reduce the depressive feelings.

This study is conducted as a randomised controlled trial with four groups. The four groups will be (1) Qigong exercise and art activity group as an integrated intervention (2) An art activity group; (3) A Qigong group; and (4) no intervention/daily activities. The investigators begins by allocating participants at random to one of the intervention groups. The process of randomising the participants will be collected by sealed-envelopes used in the selection process. The participants will assemble in one room and each participant will receive a sealed-envelope, which contains a card labelled with information regarding the intervention that will follow. The information will comprise the number of sessions, time period and checklist column that must be marked by the participants, in order to indicate that they are willing to follow the intervention. Once the participants know the intervention group that they are assigned to, the investigators will conduct an initial interview to obtain demographic information and to acquire data about the reason they decided to live in a nursing home. Finally, informed consent will be obtained from the participants during the initial interview. The intervention will be conducted in 8 weeks and consists of 16 sessions that will be given twice a week; each session will be last for 90 minutes.

Furthermore, the investigators will evaluate participants who meet the criteria before the intervention. The measurement of the inclusion and exclusion criteria will be assessed by using MMSE and the MINI Neuropsychiatric Interview. Social demographic characteristics are included to collect data about age, sex and ethnicity, education, marital status (married or never married), family group, perceived economic status (upper, middle or lower), financial resources, medical history, lifestyle/exercise habits and information relating to admission to the nursing home. The MMSE is a brief indicator of cognitive ability of the elderly, and the MINI will be used as a screening tool to measure severe psychiatric disorders. The measurements will be given before and after the intervention using WHOQOL-BREF; SWLS, BDI-II and GDS 15-item, MMSE and SF-36.

The intervention process of the social art activities will be provided and participants will use art materials, for instance, drawing paper, pencils and coloured pencils, magazine, objects, glue, scissors/box cutters, collage and additional material. The materials are selected based on the consideration that they are not too messy or too complicated to work with. The Qigong consists of nine simple and slow movements that are suitable for older people. The integrated intervention will be presented in one session; hence, Qigong will be provided as the initial therapeutic activity preceding the art activities. The healing mechanisms to depressed older people using the art activities and Qigong can be obtained during the "therapeutic process", which consists of sensory stimulation, self-exploration, self-expression, communication, understanding and explanation, symbolic thinking and creativity.

During the intervention, participants will be observed based on the observation form, to know if there is any improvement in social interaction, communication and involvement in the activities, in addition to their expression and impression during the activities. A follow-up measurement will take place 3 and 6 months after the intervention, including a follow-up interview to obtain descriptive data concerning the older person's well-being, following participation in the intervention.

The control condition consists of groups of older people engaged in regular, daily activities, for instance, watching television or just sitting and reading. The participants do activities on a regular basis in nursing homes and they are not receiving any therapeutic interventions, as above. Therefore, the investigators may consider these groups as the no-treatment groups. In addition, the participants will be assembled in one room for approximately 90 minutes and they could choose to participate in daily activities in the groups.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years or older
* Deemed to be cognitively capable of participating in an in-depth interview
* Admitted to the nursing home at least 3 months ago
* Healthy physical condition (able to walk and to do daily activity without assistance)
* Consent to randomization and follow-up.

Exclusion Criteria:

* Severe cognitive impairment or dementia based on MMSE
* Blind and have severe hearing or speech impairment that might interfere with participation in the interview
* Psychotic disorders based on MINI Neuropsychiatric Interview (Sheehan et al., 1998)
* Severe physical disorder
* Severe communication problem
* Alcohol/drug misuse.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2017-01; Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
WHOQOL-BREF | Change from Baseline to 8 weeks, 3 and 6 months
  The brief version of the World Health Organization Quality of Life (WHOQOL-BREF) (The WHO Group, 1998) was developed to assess the quality of life. It contains a total of 26 questions. All items are rated on a five-point Likert scale using response categories such as 1 represents very poor, and 5 represents very well with the statement. The instrument consists of four domains: psychological health, physiological health, social relationships, and environmental health. The test - re-test reliability for WHOQOL-BREF lies within 0.81 to 0.90.

SECONDARY OUTCOMES:
SWLS | Change from Baseline to 8 weeks, 3 and 6 months
  The satisfaction with life scale (SWLS) (Diener, 1984) was developed to assess satisfaction with the respondent's life as a whole. It consists of five statements that the client could either agree or disagree with on a scale of 1 - 7, where 1 represents strongly disagree, and 7 represents strongly agree with the statement. Diener (1985) reported a Cronbach's alpha of 0.87 for the scale and a test - retest stability coefficient of 0.82.
The Indo BDI-II | Change from Baseline to 8 weeks, 3 and 6 months
  Beck Depression Inventory-II for Indonesian general population (Beck, Steer, & Brown, 1996; Ginting, Näring, van der Veld, Srisayekti & Becker, 2013), contains 21-item self-report inventory measuring the severity of depression in adolescents and adults. All items are rated on a 4-point Likert-type scale ranging from 0 to 3, based on the severity of each item. Cronbach's alpha of the Indo BDI-II per group was .90 for healthy participants, and .91 for depressed patients. The test-retest correlation of the Indo BDI-II was significant (r = .55, p < .01).
GDS-15 | Change from Baseline to 8 weeks, 3 and 6 months
  Geriatric Depression Scale 15-item (GDS 15-item) adapted from the Sheikh and Yesavage (1986). The GDS was designed as a screening tool for depression in elderly populations. It consists of 15 questions with YES or NO answer; where YES was treated as 0 and NO-treated as 1. A score > 5 point is suggestive of depression. The Cronbach's α coefficient was 0,71.
MMSE | Change from Baseline to 8 weeks, 3 and 6 months
  Mini-Mental State Exam (MMSE; Folstein, Folstein, & McHugh, 1975) used as a brief indicator of cognitive status. It is an 11-question measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. The maximum score is 30. A score of 23 or lower is indicative of cognitive impairment.
SF-36 | Change from Baseline to 8 weeks, 3 and 6 months
  A 36-item short-form (SF-36; Ware Jr, 1993; Perwitasari, 2012) is a widely used questionnaire for measuring self-reported physical and mental health status. It is a short-form health survey with only 36 questions. Estimates of reliability in the physical and mental sections are typically above 0.90.

CONTACTS AND LOCATIONS:
Overall Officials: Roswiyani Roswiyani, M.Psi, Principal Investigator — Behavioural Science Institute, Radboud University, The Netherlands; and Tarumanagara University, Jakarta, Indonesia; Jan Spijker, Prof. dr., Study Director — Behavioural Science Institute, Radboud University, The Netherlands, and Pro Persona Mental Health Care, Depression Expertise Centre, Nijmegen, the Netherlands; Cilia Witteman, Prof. dr., Study Director — Behavioural Science Institute, Radboud University, The Netherlands
Locations (1):
- Panti wredha, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diener E. Subjective well-being. Psychol Bull. 1984 May;95(3):542-75. No abstract available. PMID 6399758
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Hays RD, Sherbourne CD, Mazel RM. The RAND 36-Item Health Survey 1.0. Health Econ. 1993 Oct;2(3):217-27. doi: 10.1002/hec.4730020305. PMID 8275167
- [Background] Thyme, K. E., Sundin, E. C., Stahlberg, G., Lindstrom, B., Eklof, H., & Wiberg, B. (2007). The outcome of short-term psychodynamic art therapy compared to short-term psychodynamic verbal therapy for depressed women. Psychoanalytic Psychotherapy, 21, 250-264.
- [Background] Wang F, Man JK, Lee EK, Wu T, Benson H, Fricchione GL, Wang W, Yeung A. The effects of qigong on anxiety, depression, and psychological well-being: a systematic review and meta-analysis. Evid Based Complement Alternat Med. 2013;2013:152738. doi: 10.1155/2013/152738. Epub 2013 Jan 14. PMID 23401706
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Ginting, H., Näring, G., van der Veld, W.M., Srisayekti, W., & Becker, E. S. (2013). Validating the Beck Depression Inventory-II in Indonesia's general population and coronary heart disease patients. International Journal of Clinical and Health Psychology, 13, 235-242. DOI: 10.1016/S1697-2600(13)70028-0.
- [Background] Sheikh, J.I., & Yesavage, J.A. (1986). Geriatric Depression Scale (GDS) recent evidence and development of a shorter version. In: Brink TL, editor. Clinical Gerontology : A Guide to Assessment and Intervention. New York: The Haworth Press, pp. 165-173.
- [Background] Ali, U. & Hasan, S. (2010). The effectiveness of relaxation therapy in the reduction of anxiety related symptoms (a case study). International Journal of Psychological Studies, 2, 2; 202-208. www.ccsenet.org/ijps
- [Background] Blomdahl, Gunnarsson, Guregård, S., & Björklund, A. (2013). A realist review of art therapy for clients with depression. The Arts in Psychotherapy, 40, 322- 330. DOI:10.1016/j.aip.2013.05.009
- [Background] Cloosterman, N.H.M., Laan, A. J., & Alphen, B.P.J.V. (2013). Characteristics of psychotherapeutic integration for depression in older adults: A delphi study. Clinical Gerontologist, 36:5, 395-410. DOI: 10.1080/07317115.2013.816815.
- [Background] Djernes JK. Prevalence and predictors of depression in populations of elderly: a review. Acta Psychiatr Scand. 2006 May;113(5):372-87. doi: 10.1111/j.1600-0447.2006.00770.x. PMID 16603029
- [Background] Etemadi, A., & Ahmadi, K. (2009). Psychological disorders of elderly home residents. Journal of Applied Sciences, 9:3, 549-554. DOI: 10.3923/jas.2009.549.554
- [Background] Gunnarsson AB, Eklund M. The Tree Theme Method as an intervention in psychosocial occupational therapy: client acceptability and outcomes. Aust Occup Ther J. 2009 Jun;56(3):167-76. doi: 10.1111/j.1440-1630.2008.00738.x. PMID 20854510
- [Background] Gunnarsson AB, Jansson JA, Eklund M. The Tree Theme Method in psychosocial occupational therapy: a case study. Scand J Occup Ther. 2006 Dec;13(4):229-40. doi: 10.1080/11038120600772908. PMID 17203673
- [Background] Hass-Cohen, N.,&Carr, R. (Eds.). (2008). Art therapy and clinical neuroscience. London, England: Jessica Kingsley.
- [Background] Isaksson, C., Norlén, A.-K., Englund, B., & Lindqvist, R. (2009). Changes in self-imagesas seen in tree paintings. The Arts in Psychotherapy, 36, 304-312. Doi:10.1016/j.aip.2009.07.004.
- [Background] Jongenelis K, Pot AM, Eisses AM, Beekman AT, Kluiter H, Ribbe MW. Prevalence and risk indicators of depression in elderly nursing home patients: the AGED study. J Affect Disord. 2004 Dec;83(2-3):135-42. doi: 10.1016/j.jad.2004.06.001. PMID 15555706
- [Background] Monti DA, Peterson C, Kunkel EJ, Hauck WW, Pequignot E, Rhodes L, Brainard GC. A randomized, controlled trial of mindfulness-based art therapy (MBAT) for women with cancer. Psychooncology. 2006 May;15(5):363-73. doi: 10.1002/pon.988. PMID 16288447
- [Background] Neufeld, E., Freeman, S., Joling, K., & Hirdes, J.P. (2014) "When the golden years are blue": Changes in depressive symptoms over time among older adults newly admitted to long-term care facilities. Clinical Gerontologist, 37:3, 298-315. DOI:10.1080/07317115.2014.885919.
- [Background] Segal, Z.V.,Williams,J.M.G.,&Teasdale,J.D.(2002). Mindfulness-based cognitive therapy for depression. New York: The Guilford Press.
- [Background] Vinson, L.D., MA , Crowther, M.R., Austin, A.D., & Guin, S.M. (2014). African Americans, mental health, and aging. Clinical Gerontologist, 37:1, 4-17. DOI: 10.1080/07317115.2013.847515.
- [Background] Beck, A. T., Steer, R. A., & Brown, G. K. (1996). Beck depression inventory-ii. San Antonio, 78(2), 490-498.
- [Background] Perwitasari, D. A. (2012). Development the validation of indonesian version of sf-36 questionnaire in cancer disease. Indonesian Journal of Pharmacy, 248-253.
- [Background] Ware, J. E. (1993). Sf-36 health survey: Manual and interpretation guide. Boston, MA: Nimrod Press.
- [Derived] Roswiyani R, Hiew CH, Witteman CLM, Satiadarma MP, Spijker J. Art activities and qigong exercise for the well-being of older adults in nursing homes in Indonesia: a randomized controlled trial. Aging Ment Health. 2020 Oct;24(10):1569-1578. doi: 10.1080/13607863.2019.1617239. Epub 2019 May 30. PMID 31146543